CLINICAL TRIAL: NCT07127900
Title: Define-PFA: Diaphragmatic Evaluation by Fluoroscopy to Identify Phrenic Nerve Dysfunction Related to Electroporation
Brief Title: Diaphragmatic Evaluation by Fluoroscopy to Identify Phrenic Nerve Dysfunction Related to Electroporation
Acronym: Define-PFA
Status: Withdrawn | Type: Observational
Why Stopped: For administrative reasons
Sponsor: Laurent Macle (Other)
Responsible Party: Sponsor-Investigator, Laurent Macle, Cardiologist electrophysiologist, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Other Study IDs: ICM-2026-3595
Record Dates: First submitted 2025-08-04; First posted 2025-08-17 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation (AF); Phrenic Nerve-related Diaphragmatic Impairment
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to better understand the potential side effects of a heart treatment called PFA (Pulsed Field Ablation), used to treat an arrhythmia known as atrial fibrillation. This technique has already been in clinical use for several years.

The goal of the study is to detect a possible adverse effect of this procedure: injury to the phrenic nerve, which could result in paralysis of one side of the diaphragm. The diaphragm is an important muscle for breathing and can occasionally be affected during certain cardiac ablation procedures.

To assess this, patients will undergo a dynamic chest X-ray (fluoroscopy) before and after the procedure. If diaphragm movement appears reduced afterward, a follow-up exam will be performed at 3 months to monitor the evolution. Patients presenting with a fluoroscopic abnormality at Month 3 will undergo a follow-up at Month 6. If the abnormality persists at M6, follow-up will be extended to Month 12.

The study does not involve any experimental treatment or changes to standard medical care, and there are no additional risks associated with the planned exams. It is entirely observational. All data will be used anonymously to help improve the safety of current techniques.

DETAILED DESCRIPTION:
Study Type This is a prospective, observational, multicenter study conducted in four electrophysiology centers. The study does not involve any experimental intervention or modification of standard care. It is based on the systematic observation of a complementary imaging exam (dynamic fluoroscopy) performed before and after a PFA procedure, as part of the routine management of atrial fibrillation.

Participation Duration

The maximum duration of participation for each patient is twelve (12) months. Follow-up includes:

an inclusion visit with pre-procedure fluoroscopy,

a post-procedure fluoroscopy performed before hospital discharge (on the day of the procedure or the following day, depending on local practices),

a 3-6 and 12 month visit with fluoroscopy, only if an abnormality was detected in the post-procedure assessment.

General Methodology The study aims to include 250 consecutive patients undergoing PFA for atrial fibrillation, regardless of the single-shot system used (FARAPULSE™, PULSE SELECT™, VARIPULSE™, or VOLT™), at the discretion of each operator.

Dynamic fluoroscopy will be performed before the catheter ablation using a PFA system, and repeated afterward before the patient's discharge-on the same day or the following day, depending on the center's practice. The images will be stored and analyzed to assess diaphragmatic excursion (in millimeters). Exams will be considered of sufficient quality if the excursion of at least one hemidiaphragm is ≥35 mm, and optimal if ≥40 mm. Diaphragmatic impairment will be defined as an asymmetry ≥15% in cranio-caudal excursion between hemidiaphragms after the procedure. Patients with diaphragmatic impairment will be invited for a follow-up fluoroscopy at three months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paroxysmal or persistent atrial fibrillation (AF), documented by any method: ECG, Holter, invasive monitoring (implantable device memory), or non-invasive monitoring (connected devices).
* Ablation indication decided as part of routine care, according to society guidelines.
* First ablation procedure (including pulmonary vein isolation) planned using a commercially available PFA catheter.
* Ability to perform diaphragmatic fluoroscopic evaluation before and after the procedure (before hospital discharge).

Exclusion Criteria:

* Patients presenting with one or more of the following conditions will be excluded from the study:
* Known history of diaphragmatic paralysis (right-sided or bilateral) or preexisting clinical suspicion.
* History of atrial fibrillation ablation.
* History of neuromuscular disease.
* History of major thoracic surgery or chronic pulmonary pathology likely to impair diaphragmatic motion.
* Diaphragmatic paralysis diagnosed during the pre-procedure fluoroscopic assessment.
* Inability to perform post-procedure fluoroscopic control (due to logistical limitations, patient refusal, or contraindication to radiation exposure).
* Current pregnancy or breastfeeding.
* Concurrent participation in another interventional study that may interfere with the objectives of the present research.
* Significant cognitive impairment or inability to understand the study objectives or provide valid consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study plans to include 250 consecutive patients undergoing atrial fibrillation ablation by PFA, regardless of the "one-shot" system used (FARAPULSE™, PULSE SELECT™, VARIPULSE™, or VOLT™), at the discretion of each operator.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of diaphragmatic abnormality | Hospital discharge
  asymmetry ≥ 15%, paradoxical excursion

SECONDARY OUTCOMES:
Respiratory symptoms associated with diaphragmatic paralysis | Hospital discharge: up to 48hrs post-procedure
  dyspnea, inspiratory discomfort, reduced physical capacity
Correlation between technical characteristics of the ablation and the occurrence of diaphragmatic paralysis. | Hospital discharge: up to 48hrs post-procedure
  in particular, the type of catheter used
Final status of the recovery of diaphragmatic abnormalities | 12 months post-procedure
  complete recovery / partial recovery / no recovery of diaphragmatic abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Macle, MD, Principal Investigator — Montreal Heart Institute - Montréal, QC; Frederic Franceschi, MD. Pr., Principal Investigator — Auckland City Hospital (ACH)

IPD SHARING:
Plan to Share IPD: No